CLINICAL TRIAL: NCT01270867
Title: Thrombectomy REvascularization of Large Vessel Occlusions in Acute Ischemic Stroke (TREVO 2)
Brief Title: Randomized Trial Evaluating Performance of the Trevo Retriever Versus the Merci Retriever in Acute Ischemic Stroke
Acronym: TREVO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DQR0038
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemia; Stroke; Ischemic Stroke; Mechanical Thrombectomy; Brain; Brain clot; Cerebrovascular disease; Recanalization; Revascularization
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Merci Retriever (Active Comparator): Merci Retriever is the predicate product that received FDA clearance in 2004. Merci Retriever a first generation mechanical thrombectomy device intended to remove clot and restore blood flow in a neurovascular vessel in the setting of acute ischemic stroke.
  Interventions: Device: Mechanical Thrombectomy
- Trevo Stentriever (Experimental): Trevo Retriever is a second generation mechanical thrombectomy device intended to remove clot and restore blood flow in a neurovascular vessel in the setting of acute ischemic stroke. The Trevo Retriever is a type of stent, specifically design to allow for clot integration into the device. The clot in the retriever is then removed and blood flow is restored.
  Interventions: Device: Mechanical Thrombectomy

INTERVENTIONS:
Device: Mechanical Thrombectomy — Each arm will use either Merci or Trevo as the primary Mechanical Thrombectomy device.

SUMMARY:
To determine if the Trevo Retriever is as good or better than the Merci Retriever in restoring blood flow to the brain of a patient experiencing an acute ischemic stroke in a large vessel.

DETAILED DESCRIPTION:
The TREVO 2 protocol was designed to assess the safety and effectiveness of the Trevo Retriever device and determine if it is substantially equivalent to the predicate Merci Retriever. The trial utilized a Primary Effectiveness Endpoint of revascularization and a composite Primary Safety Endpoint that included procedure-related serious adverse events occurring within 24 hours of the procedure. Subjects who presented to enrolling centers with large ischemic strokes were screened for eligibility in the study. If a subject met eligibility criteria, then Informed Consent was obtained prior to commencing the angiogram. If all inclusion/exclusion criteria were confirmed, including the angiographic criteria, then the subject was randomized.The Primary Effectiveness Endpoint was successful revascularization of the target occlusion, using the TICI score. Success was determined by the central Core Lab.The Primary Safety Endpoint is a composite endpoint, described in the protocol as the "Incidence of procedure-related serious adverse events (PRSAEs) through 24 hours post procedure (-6/+12 hours) defined as: vascular perforation or intramural arterial dissection, symptomatic ICH, embolization to a previously uninvolved territory, access site complication requiring surgical repair or blood transfusion, intra-procedural mortality, device failure (in vivo breakage), or any other complications judged by the Clinical Events Committee (CEC) to be related to the procedure."

ELIGIBILITY:
Key Inclusion Criteria:

* Patient presenting with clinical signs and symptoms consistent with a diagnosis of Acute Ischemic Stroke, and:

  * Patient has failed IV t-PA therapy Or
  * Patient is contraindicated for IV t-PA administration
* NIHSS 8 < NIHSS < 29
* Anticipated life expectancy of at least 6 months
* No significant pre-stroke disability (mRS < 1)
* Written informed consent to participate given by patient or legal representative
* Angiographic confirmation of a persistent large vessel occlusion in the internal carotid, middle cerebral (M1 and/or M2 segments), basilar and/or vertebral arteries
* Treatable within 8 hours of symptom onset, defined as the first pass being made with the assigned study device

Key Exclusion Criteria:

* Abnormal blood pressure and/or blood coagulation lab values
* Pregnancy
* Patient participating in another investigational drug or device study
* More than 1/3 of MCA or equivalent in non-MCA territory
* Baseline evidence of significant mass effect with midline shift, or hemorrhage, or intracranial tumor
* Bilateral stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — Emory University; Helmi Lutsep, MD, Principal Investigator — Oregon Health and Science University; Wade Smith, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States

REFERENCES:
- [Result] Nogueira RG, Lutsep HL, Gupta R, Jovin TG, Albers GW, Walker GA, Liebeskind DS, Smith WS; TREVO 2 Trialists. Trevo versus Merci retrievers for thrombectomy revascularisation of large vessel occlusions in acute ischaemic stroke (TREVO 2): a randomised trial. Lancet. 2012 Oct 6;380(9849):1231-40. doi: 10.1016/S0140-6736(12)61299-9. Epub 2012 Aug 26. PMID 22932714
- [Derived] Winningham MJ, Haussen DC, Nogueira RG, Liebeskind DS, Smith WS, Lutsep HL, Jovin TG, Xiang B, Nahab F. Periprocedural heparin use in acute ischemic stroke endovascular therapy: the TREVO 2 trial. J Neurointerv Surg. 2018 Jul;10(7):611-614. doi: 10.1136/neurintsurg-2017-013441. Epub 2017 Oct 31. PMID 29089415
- [Derived] Shi ZS, Liebeskind DS, Xiang B, Ge SG, Feng L, Albers GW, Budzik R, Devlin T, Gupta R, Jansen O, Jovin TG, Killer-Oberpfalzer M, Lutsep HL, Macho J, Nogueira RG, Rymer M, Smith WS, Wahlgren N, Duckwiler GR; Multi MERCI, TREVO, and TREVO 2 Investigators. Predictors of functional dependence despite successful revascularization in large-vessel occlusion strokes. Stroke. 2014 Jul;45(7):1977-84. doi: 10.1161/STROKEAHA.114.005603. Epub 2014 May 29. PMID 24876082
- See also: Concentric Medical Website — http://www.concentric-medical.com
- See also: American Stroke Association — http://www.strokeassociation.org/STROKEORG/

RESULTS

PARTICIPANT FLOW:
Groups:
- Merci Retriever: Patients who were randomized to the Merci Retriever
- Trevo Stentriever: Patients who were randomized to the Trevo Stentriever
Period: Overall Study
Arm/Group | Merci Retriever | Trevo Stentriever
Started | 90 | 88
Completed | 89 | 88
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Merci Retriever | Trevo Stentriever | Total
Number analyzed (Participants) | 90 | 88 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (14.7) | 67.4 (13.9) | 67.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 102
  Male | 36 | 40 | 76
Region of Enrollment [Number; unit: participants]
  United States | 89 | 88 | 177
  Spain | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint
Description: Revascularization of the occluded territory, defined as at least TICI 2 flow in the treated territory after use of the assigned device.
  Thrombolysis in Cerebral Infarction (TICI) grading system for perfusion (ie blood flow through a vessel) Grade 0:No Perfusion. No antegrade flow beyond the point of occlusion. Grade 1:Penetration With Minimal Perfusion. Grade 2:Partial Perfusion. Grade 2a:Only partial filling (<2/3) of the entire vascular territory is visualized.
  Grade 2b:Complete filling of all of the expected vascular territory is visualized, but slower ...
  Grade 3:Complete Perfusion. For complete info see Higashida RT, Furlan AJ, Roberts H, Tomsick T, Connors B et al. (2003) Trial design and reporting standards for intra-arterial cerebral thrombolysis for acute ischemic stroke. Stroke 34: e109-e137.10.1161/01.STR.0000082721.62796.09 PubMed: 12869717[PubMed]
Time Frame: acute/procedural
Population: Intent to treat analysis was performed. The non-inferiority hypothesis was tested with Blackwelder's method, assuming a one-sided alpha=0.025 and a clinically relevant non-inferiority margin of 10%.
Measure: Number; unit: participants
Groups:
- Merci Retriever: Patients who were randomized to receive the Merci Retriever.
- Trevo Stentriever: Patients who were randomized to receive the Trevo Stentriever.
Arm/Group | Merci Retriever | Trevo Stentriever
Number analyzed (Participants) | 90 | 88
participants | 54 | 76

2. Primary Outcome: Primary Safety Endpoint
Description: Incidence of procedure-related serious adverse events (PRSAEs) through 24 hours post procedure (-6/+12 hours).
Time Frame: within 24 hours of procedure
Measure: Number; unit: participants
Arm/Group | Merci Retriever | Trevo Stentriever
Number analyzed (Participants) | 90 | 88
participants | 21 | 13

3. Secondary Outcome: Secondary Endpoint
Description: Good clinical outcomes at 90 days, as assessed by mRS (a "good" clinical outcome is defined as mRS </= 2)
  mRS 0-2 indicates functional independence 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead. https://en.wikipedia.org/wiki/Modified_Rankin_Sca
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Merci Retriever | Trevo Stentriever
Number analyzed (Participants) | 87 | 85
participants | 19 | 34

4. Secondary Outcome: Secondary Endpoint
Description: All cause mortality at 90 days
Time Frame: procedure through 90 days
Measure: Number; unit: participants
Arm/Group | Merci Retriever | Trevo Stentriever
Number analyzed (Participants) | 89 | 88
participants | 21 | 29

5. Secondary Outcome: Secondary Endpoint
Description: Incidence of asymptomatic intracranial hemorrhages (ICH) within 24 (-6/+12) hours post procedure
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Merci Retriever | Trevo Stentriever
Number analyzed (Participants) | 90 | 88
participants | 48 | 36

ADVERSE EVENTS:
Time Frame: Each subject was followed for 90 days; The study period was 1 year.
Description: A study specific AE classification system was used to categorize Site Reported AEs and SAEs.
  The study used an independent clinical events committee, CT and MRI imaging core laboratory, a separate angiography core laboratory, and an independent data safety and monitoring board (DSMB) to ensure appropriate oversight and analysis.
Arm/Group | Merci Retriever | Trevo Stentriever
Serious Adverse Events (participants affected / at risk) | 39/90 | 41/88
Other Adverse Events (participants affected / at risk) | 73/90 | 71/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Merci Retriever (N=90) | Trevo Stentriever (N=88)
Acute Mental Status Change/Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Edema (Nervous system disorders) | 8 (8) | 10 (11)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Difficulty Swallowing) (Nervous system disorders) | 4 (4) | 1 (1)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
IVH (Nervous system disorders) | 0 (0) | 1 (1)
SAH (Nervous system disorders) | 5 (5) | 3 (3)
ICH - HI -1 (Nervous system disorders) | 4 (4) | 0 (0)
ICH - HI -2 (Nervous system disorders) | 1 (1) | 1 (1)
ICH - PH1 (Nervous system disorders) | 5 (5) | 5 (5)
ICH - PH2 (Nervous system disorders) | 3 (3) | 3 (3)
Neurologic Decline (Nervous system disorders) | 2 (2) | 5 (5)
New Ischemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Late ICH (Nervous system disorders) | 2 (2) | 2 (2)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Progression of index Stroke (Nervous system disorders) | 6 (6) | 8 (8)
Reocclusion at the site of original occlusion or proximal to original occlusion (Vascular disorders) | 1 (1) | 0 (0)
Seizure - New Onset (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsiveness (Nervous system disorders) | 0 (0) | 1 (1)
Arrhythmia - Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 1 (1)
Hypotension - Sustained - Tx (Cardiac disorders) | 1 (1) | 2 (2)
Stress Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Other (Gastrointestinal disorders) | 1 (1) | 0 (0)
Occult Blood (Gastrointestinal disorders) | 1 (1) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Joint/Extremity Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Access Site Complication (Surgical and medical procedures) | 0 (0) | 2 (2)
Intramural Arterial Dissection (Surgical and medical procedures) | 1 (1) | 0 (0)
Hemoptysis (bloody sputum) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Respiratory Failure - Acute (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 (1) | 3 (3)
Drug Reaction (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Positive Cultures (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Events With an Outcome of Death (General disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Merci Retriever (N=90) | Trevo Stentriever (N=88)
Cerebral Edema (Nervous system disorders) | 8 (8) | 4 (4)
Headache (Nervous system disorders) | 8 (8) | 8 (9)
Dysphagia (Difficulty Swallowing) (Nervous system disorders) | 20 (20) | 14 (14)
SAH (Nervous system disorders) | 8 (8) | 1 (1)
ICH - HI -1 (Nervous system disorders) | 7 (7) | 7 (7)
ICH - PH1 (Nervous system disorders) | 8 (8) | 4 (4)
Neurologic Decline (Nervous system disorders) | 6 (6) | 0 (0)
Arrhythmia - Tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 9 (9)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea and Vomiting (Non-Neuro) (Gastrointestinal disorders) | 3 (3) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 17 (17) | 14 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10) | 8 (8)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 24 (32) | 15 (22)
Joint/Extremity Pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 9 (10)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Respiratory Failure - Acute (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 12 (12) | 9 (10)
Fever (General disorders) | 5 (5) | 4 (4)
Positive Cultures (General disorders) | 7 (7) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 18 (19) | 14 (15)
Hematuria (Renal and urinary disorders) | 1 (2) | 6 (6)
Urinary Retention (Renal and urinary disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days